CLINICAL TRIAL: NCT07268924
Title: The Effect of Propofol Versus Lidocaine on Emergence Agitation in Children Undergoing Tonsillectomy.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hesham Bahaa-eldin Mohamed, Resident doctor at anesthesia & ICU depatrtment, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EA-CHT-PvL-2025
Record Dates: First submitted 2025-09-24; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Emergence Delirium, Anesthesia
Keywords: Emergence agitation in anesthesia
MeSH Terms: conditions — Emergence Delirium | interventions — Propofol

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group ( p ) recieve 1mg /kg of propofol (Active Comparator)
  Interventions: Drug: Propofol
- Group ( L ) recieve 1.5 mg/kg of lidocaine (Active Comparator)
  Interventions: Drug: Lidocaine %2 ampoule

INTERVENTIONS:
Drug: Propofol — In pediatric tonsillectomy after the end of surgery, patient will recieve 1 mg/kg of propofol iv bolus
  Arms: Group ( p ) recieve 1mg /kg of propofol
Drug: Lidocaine %2 ampoule — In pediatric tonsillectomy after the end of the surgery , patient will recieve 1.5 mg/kg of lidocaine iv bolus
  Arms: Group ( L ) recieve 1.5 mg/kg of lidocaine

SUMMARY:
This study aim to compare the effect of intravenous propofol versus intravenous lidocaine on emergence agitation in children undergoing tonsillectomy or adenotonsillectomy under general anesthesia.

DETAILED DESCRIPTION:
Tonsillectomy is one of the common surgeries in children, which is associated with many morbidities such as postoperative pain, nausea, vomiting, bleeding, dehydration and emergence agitation .

Emergence agitation (EA) is a prevalent occurance following sevoflorane anesthesia , with an incidence of up to 80% , particularly among preschool children EA is characterised by a dissociated state of consciousness' in which the child displays irritability, anxiety , and inconsolable crying, kicking, or thrashing behavior Furthermore , EA in children can potentially be dangerous as it may lead to incidents such as falling out of bed , removal of surgical dressings , intravenous catheters , increase stress for healthcare providera and parents , higher costs due to prolonged recovery stay .³ The mechanism of EA remains unclear. The proposed risk factors of EA include age ,preoperative anxiety,, type of surgery, emergency operation, use of inhalational anesthetics , long duration of surgery.

Several pharmacological prophylactic interventions ,including opioids analgesics , benzodiazepines, α2-adrenergic receptor agonists such as clonidine , have been studied for their potential to reduce incedence of EA .

Propofol, short acting intravenous anesthetic, is known for smoother emergence and sedative properties. Lidocaine, administered intravenously, has analgesic, anti-inflammatory, and sedative effects. There is limited direct comparison between these two drugs specifically in pediatrc tonsillectomy with EA.

So, does intravenous lidocaine compared with propofol reduce the incidence and severity of emergence agitation in children undergoing tonsillectomy or adenotonsillectomy ?

ELIGIBILITY:
Inclusion Criteria:

* Elective tonsillectomy operation
* pediaterics between ( 4 : 7 ) years old
* ASA I OR II

Exclusion Criteria:

* emergency cases as bleeding tonsills
* ASA III OR IV

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To compare the incidence and severity of emergence agitation (EA) between children receiving propofol and those receiving lidocaine using Pediatric Anesthesia Emergence Delirium (PAED) scale. | Within 30 minutes after extubation
  Pediatric Anesthesia Emergence Delirium (PAED) scale (range 0-20; higher scores indicate more severe agitation).
To compare the incidence and severity of emergence agitation (EA) between children receiving propofol and those receiving lidocaine using WATCHA scale | Within 30 minutes after extubation.
  Watcha agitation scale (range 0-4; higher scores indicate more severe agitation).

SECONDARY OUTCOMES:
emergence time from anesthesia | Within 30 minutes after extubation.
peaked PAED scores | Within 30 minutes after extubation.
  Pediatric Anesthesia Emergence Delirium (PAED) scale (range 0-20; higher scores indicate more severe agitation).
extubation time | Within 30 minutes after extubation.
post-operative pain using FLACC score | Within 30 minutes after extubation.
  The FLACC scale is used to assess postoperative pain in children. It consists of 5 categories (Face, Legs, Activity, Cry, Consolability), each scored 0-2, giving a total score range of 0-10.
Hemodynamic effects as hypotention and bradycardia | Within 30 minutes after extubation.
Post operative nausea and vomitting | Within 30 minutes after extubation.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Ahmed SA, Omara AF. The Effect of Glossopharyngeal Nerve Block on Post-Tonsillectomy Pain of Children; Randomized Controlled Trial. Anesth Pain Med. 2019 Apr 30;9(2):e90854. doi: 10.5812/aapm.90854. eCollection 2019 Apr. PMID 31341828
- [Result] Ji JY, Park JS, Kim JE, Kim DH, Chung JH, Chun HR, Jung HS, Yoo SH. Effect of esmolol and lidocaine on agitation in awake phase of anesthesia among children: a double-blind, randomized clinical study. Chin Med J (Engl). 2019 Apr 5;132(7):757-764. doi: 10.1097/CM9.0000000000000141. PMID 30741832
- [Result] Manouchehrian N, Jiryaee N, Moheb FA. Propofol versus lidocaine on prevention of laryngospasm in tonsillectomy: A randomized clinical trial. Eur J Transl Myol. 2022 Jun 29;32(3):10581. doi: 10.4081/ejtm.2022.10581. PMID 35766592
- [Result] Watcha MF, Ramirez-Ruiz M, White PF, Jones MB, Lagueruela RG, Terkonda RP. Perioperative effects of oral ketorolac and acetaminophen in children undergoing bilateral myringotomy. Can J Anaesth. 1992 Sep;39(7):649-54. doi: 10.1007/BF03008224. PMID 1394752
- [Result] Sikich N, Lerman J. Development and psychometric evaluation of the pediatric anesthesia emergence delirium scale. Anesthesiology. 2004 May;100(5):1138-45. doi: 10.1097/00000542-200405000-00015. PMID 15114210
- [Result] Clivio S, Putzu A, Tramer MR. Intravenous Lidocaine for the Prevention of Cough: Systematic Review and Meta-analysis of Randomized Controlled Trials. Anesth Analg. 2019 Nov;129(5):1249-1255. doi: 10.1213/ANE.0000000000003699. PMID 30169416
- [Result] Mokhtar AM, Badawy AA. [Low dose propofol vs. lidocaine for relief of resistant post-extubation laryngospasm in the obstetric patient]. Braz J Anesthesiol. 2018 Jan-Feb;68(1):57-61. doi: 10.1016/j.bjan.2017.03.009. Epub 2017 Jul 25. PMID 28754225
- [Result] Malviya S, Voepel-Lewis T, Ramamurthi RJ, Burke C, Tait AR. Clonidine for the prevention of emergence agitation in young children: efficacy and recovery profile. Paediatr Anaesth. 2006 May;16(5):554-9. doi: 10.1111/j.1460-9592.2006.01818.x. PMID 16677266
- [Result] Na HS, Song IA, Hwang JW, Do SH, Oh AY. Emergence agitation in children undergoing adenotonsillectomy: a comparison of sevoflurane vs. sevoflurane-remifentanil administration. Acta Anaesthesiol Scand. 2013 Jan;57(1):100-5. doi: 10.1111/aas.12006. Epub 2012 Oct 30. PMID 23110746
- [Result] Kanaya A. Emergence agitation in children: risk factors, prevention, and treatment. J Anesth. 2016 Apr;30(2):261-7. doi: 10.1007/s00540-015-2098-5. Epub 2015 Nov 24. PMID 26601849
- [Result] Acar HV, Yilmaz A, Demir G, Eruyar SG, Dikmen B. Capsicum plasters on acupoints decrease the incidence of emergence agitation in pediatric patients. Paediatr Anaesth. 2012 Nov;22(11):1105-9. doi: 10.1111/j.1460-9592.2012.03876.x. PMID 22553919
- [Result] Chen J, Shi X, Hu W, Lin R, Meng L, Liang C, Ma X, Xu L. Comparing different administration methods of subanaesthetic propofol to mitigate emergence agitation in preschool children undergoing day surgery: a double-blind, randomised controlled study. BMJ Paediatr Open. 2025 Mar 15;9(1):e002376. doi: 10.1136/bmjpo-2023-002376. PMID 40090678
- [Result] Xie M, Li XK, Peng Y. Magnesium sulfate for postoperative complications in children undergoing tonsillectomies: a systematic review and meta-analysis. J Evid Based Med. 2017 Feb;10(1):16-25. doi: 10.1111/jebm.12230. PMID 27787936
- [Result] Stalfors J, Ericsson E, Hemlin C, Hultcrantz E, Mansson I, Roos K, Hessen Soderman AC. Tonsil surgery efficiently relieves symptoms: analysis of 54 696 patients in the National Tonsil Surgery Register in Sweden. Acta Otolaryngol. 2012 May;132(5):533-9. doi: 10.3109/00016489.2011.644252. Epub 2012 Jan 11. PMID 22235871